CLINICAL TRIAL: NCT03715075
Title: Intra-epidermal Nerve Fibre Density and Its Relationship to Post-caesarean Section Pain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal Infirmary of Edinburgh (Other)
Responsible Party: Principal Investigator, Oliver Daly, Consultant Anaesthetist, NRS Career Research Fellow, Royal Infirmary of Edinburgh
Other Study IDs: IENFD in Caesarean Section
Record Dates: First submitted 2018-10-10; First posted 2018-10-22 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Chronic Pain; Cesarean Section Complications
Keywords: Intra-epidermal; nerve fibre density
MeSH Terms: conditions — Chronic Pain | interventions — Cesarean Section

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Post-caesarean section group: This single cohort observational study shall recruit women undergoing elective caesarean section within the Simpson's Centre for Reproductive Health (SCRH).
  Interventions: Procedure: Caesarean Section

INTERVENTIONS:
Procedure: Caesarean Section — Caesarean Section

SUMMARY:
Chronic pain is a significant burden to the individual and society with post-surgical pain identified as a research priority for the speciality of anaesthesia.

The objectives are to explore the relationship between IENFD and pain after caesarean section and to explore the characteristics of post-caesarean section pain.

The hypothesis is that reduced pre-operative IENFD at the surgical site will correlate with risk of developing CPSP.

DETAILED DESCRIPTION:
Based on the existing evidence, chronic pain after caesarean section appears to have an incidence between 12-18%; with the current Scottish caesarean section rate, this equates to approximately 3000 young, active women each year. Their lives may be affected by pain leading to increased analgesic use, a restriction of daily activities, decreased quality of life, and increased utilisation of healthcare services. The National Institute of Academic Anaesthesia (NIAA) has undertaken a priority setting exercise with 1700 patients and clinicians and declared the prevention of chronic post-surgical pain as one of its top 10 research priorities for the speciality of Anaesthesia.

IENFD is calculated by counting the number of nerve fibres crossing the basement membrane through direct visualisation of a skin biopsy that has undergone immunohistochemical staining. Skin biopsy is minimally invasive and allows visualisation of small fibre nociceptors that are not suitable for identification or study through nerve conduction studies.

There is emerging evidence from clinical studies that chemotherapy induced peripheral neuropathy (CIPN) patients have altered sensory innervation compared to healthy controls. In both colorectal cancer and multiple myeloma, pre-oncological treatment reductions in IENFD were associated with changes in physical testing, confirming a subclinical sensory deficit. The degree of loss of IENFD correlates with development of mechanical hyperalgesia and patients with greater sensory loss at baseline developed more symptoms during and after chemotherapy. To date there have been no studies that have examined the relationship between a patient's pre-operative IENFD and the development of chronic post-surgical pain.

This single cohort observational study shall recruit women undergoing elective caesarean section within the Simpson's Centre for Reproductive Health (SCRH). All women shall be sent a patient information sheet with a covering letter one week prior to the date of the surgery.

There shall be five discrete data collection points:

* Before caesarean section: a researcher shall collect patient demographic data, information about their general health and ask the patient to complete a Hospital Anxiety & Depression Scale (HADS).
* At the time of caesarean section: a punch biopsy shall be taken from the incision site and be sent for INEFD testing. This will be carried out once surgical anaesthesia has been achieved thereby not causing any discomfort to the participant.
* 24 hours post caesarean section: The patient's electronic record shall be consulted, if there has been any traumatic events (e.g. death or significant injury to the baby) then we shall remove the patient from the study to prevent causing any further emotional distress. The participant will be informed of this.

A researcher shall ask the patient to complete the BPI (omitting section 9 that is non-applicable).

• 3 & 6 months post caesarean section: The patient's electronic record shall be consulted, if there has been any traumatic events (e.g. death or significant injury to the baby) then we shall remove the patient from the study to prevent causing any further emotional distress. The participant will be informed of this.

A researcher shall contact participants by phone and, if they have pain, ask them to complete the following questionnaires: HADS, BPI and S-LANSS.

A researcher shall attempt to contact the patient twice via telephone, leaving a message if able, but if there is no answer or response then an assumption will be made that the participant wishes to longer be involved. No further attempts at contact will be made.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing an elective caesarean section
* Aged 18-65 years

Exclusion Criteria:

* Women undergoing urgent caesarean section
* Women with little or no English language skills - the questionnaires used are only validated for use in the English language.
* Women with cognitive impairment or mental health disorder that inhibits their ability to provide consent and/or participate in follow-up

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women undergoing an elective caesarean section
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-07-01 (Estimated); Study Completion 2019-07-01 (Estimated)

PRIMARY OUTCOMES:
Chronic Pain | 6 months
  Does the patient have pain at the operation site. A binary measure (yes or no).

SECONDARY OUTCOMES:
Brief Pain Inventory Score | 6 months
  For those with pain at 6 months, a BPI score will be recorded. The total score gives a measure of pain intensity and impact on function.
Short Leeds Assessment of Neuropathic Signs and Symptoms | 6 months
  For those with pain at 6 months, an S-LANSS score will be recorded. A total score >12 suggests that pain is of a neuropathic origin.

CONTACTS AND LOCATIONS:
Locations (1):
- Oliver Daly, Edinburgh, Midlothian, United Kingdom

IPD SHARING:
Plan to Share IPD: No